CLINICAL TRIAL: NCT06221319
Title: EFFECT OF SACRAL ERECTOR SPINA PLAN BLOCK ON RECOVERY QUALITY AFTER TOTAL HIP ARTHROPLASTY
Brief Title: EFFECT OF SACRAL ERECTOR SPINA PLAN BLOCK ON TOTAL HIP ARTHROPLASTY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Konya City Hospital (Other)
Responsible Party: Principal Investigator, Muhammed Halit Satici, Specialist, the member of the Department of Anesthesiology, Konya City Hospital, M.D, Konya City Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: total hıp arthroplasty
Record Dates: First submitted 2023-12-11; First posted 2024-01-24 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Postoperative Pain
Keywords: pain; interfascial plan block.
MeSH Terms: conditions — Pain, Postoperative; Pain

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (No Intervention): Group K IV to patients paracetamol 1 gr. It will be administered 3x1 + Dexketoprofen 50 mg 2x1. All patients will be administered 1mg/kg tramadol as rescue analgesic when NRS is 3 and above . 4mg IV to all patients with nausea and vomiting Ondansetron will be administered.
- Sacral erektör spinae plane group (Active Comparator): sacral erector spinae plane will be applied to patients in Group S
  Interventions: Other: sacral erectör spinae plane group

INTERVENTIONS:
Other: sacral erectör spinae plane group — sacral erectör spinae plane will be applied to patients in Group S
  Arms: Sacral erektör spinae plane group

SUMMARY:
Total hip arthroplasty (THA) is a surgery that relieves hip joint pain and improves its functions and is widely performed in the elderly population. New analgesic methods need to be developed to protect these patients from the pain and side effects of opioids used for treatment. Many scales are available to indicate postoperative patient recovery. One of these is the quality of recovery-15 (QoR-15) recovery test, which was first applied by Stark et al. in 2013. We think that an ESPB applied from the sacral region will spread to the lumbar region by diffusion, affect the lumbar plexus, and provide complete analgesia in the ventral and dorsal regions of the hip by affecting the sacral plexus in the sacral region. The investigator's primary aim in this study is to evaluate the effect of sacral erector spinae plane block (S-ESPB) on the quality of recovery and healing after TKA through the QoR-15 score and to evaluate its effect on postoperative pain.

DETAILED DESCRIPTION:
Total hip arthroplasty (THA) is a surgery that relieves hip joint pain and improves its functions and is widely performed in the elderly population. New analgesic methods need to be developed to protect these patients from the pain and side effects of opioids used for treatment. Many scales are available to indicate postoperative patient recovery. One of these is the quality of recovery-15 (QoR-15) recovery test, which was first applied by Stark et al. in 2013. The investigators think that an ESPB applied from the sacral region will spread to the lumbar region by diffusion, affect the lumbar plexus, and provide complete analgesia in the ventral and dorsal regions of the hip by affecting the sacral plexus in the sacral region. The investigator's primary aim in this study is to evaluate the effect of sacral erector spinae plane block (S-ESPB) on the quality of recovery and healing after TKA, through the QoR-15 score, and to evaluate its effect on postoperative pain.

Anesthesia Technique and Analgesia Protocol a standard to measure postoperative pain severity after THA, and intravenous injection is used as a standard in patients with no contraindications within the scope of the multimodal analgesia protocol. paracetamol 1 gr. 3x1 + Dexketoprofen 50 mg 2x1 and when NRS is 3 and above, 1mg/kg tramadol is administered as a rescue analgesic. In addition, ESPB is applied to patients as a part of multimodal analgesia after THA surgery, unless there are contraindications in the hospitals where the study will be conducted. And 4 mg IV is routinely administered to patients with postoperative nausea and vomiting. Ondansetron is administered . All patients will receive routine monitoring and routine anesthesia management. 20 gauge to patients Intravenous ( IV ) cannulation is provided and 15ml/kg/ h Isotonic fluid will be started. The spinal anesthesia will be applied to the patients by administering 3cc of 0.5% bupivacaine through the L3-L4 or L4-L5 intervertebral space. Patients will then be released to the surgical team for THA surgery. After the surgical procedure is completed, patients will be transferred to the postanesthetic care unit (PACU) for observation. S-ESPB will be applied to patients in Group S

ELIGIBILITY:
Inclusion Criteria:

* Patients who will undergo unilateral THA
* Spinal anesthesia
* 18-80-year-old patients
* Patients with ASA I-IV
* Patients who will stay in the hospital for at least 24 hours

Exclusion Criteria:

* Patients who do not want to give consent
* Patients under 18 years of age and over 80 years of age
* Patients for whom regional anesthesia is contraindicated
* Patients with confusion
* Patients with ASA V and above
* Patients with abnormal bleeding profile
* Patients using anticoagulants
* Patients with infection in the area to be treated
* Emergency cases

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2024-01-24 (Actual); Primary Completion 2024-04-15 (Actual); Study Completion 2024-04-15 (Actual)

PRIMARY OUTCOMES:
Quality of recovery-15T | One day
  The primary evaluation criteria will be the recording of QoR -15 scores, which indicate the quality of recovery of patients before and at 24 hours after surgery .

CONTACTS AND LOCATIONS:
Locations (1):
- Konya City Hospital, Konya, Turkey (Türkiye)